CLINICAL TRIAL: NCT07116304
Title: Comparative Efficacy of Intravenous Parecoxib Versus Lidocaine in Reducing Propofol Injection Pain: A Randomized Controlled Trial
Brief Title: Comparative Efficacy of IV Parecoxib vs Lidocaine in Reducing Propofol Injection Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Mohammed Hamood Alrashdi, Resident Doctor, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCMSS-MREC 023/2025
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Preventing Propofol Pain on Injection
Keywords: randomised controlled trial; parecoxib; propofol; NSAIDs; pain on injection
MeSH Terms: interventions — Lidocaine; parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parecoxib (Active Comparator): Patients in this group will receive IV parecoxib 40 mg (the standard full dose for an adult) diluted to a total volume of 5 mL with normal saline. The study drug will be injected into the IV cannula on the dorsum of hand **with a tourniquet applied** on the mid-arm (upper forearm) to occlude venous return. The tourniquet (elastic band) pressure will be just enough to distend veins (similar to when drawing blood) but not cause excessive discomfort. The parecoxib solution will be given over ~5-10 seconds. The tourniquet will remain in place for **2 minutes** after injection, then released. This technique of venous occlusion is borrowed from Bier block and previous studies, aiming to localize the drug in the vein for a short period to maximize local effect. then propofol will be administered.
  Interventions: Drug: Parecoxib 40mg
- Lidocaine (Active Comparator): Patients in this group will receive IV lidocaine at a dose of 0.5 mg/kg (ideal body weight) up to a maximum of 50 mg, diluted to a total of 5 mL. The lidocaine will be given into the hand IV cannula **with a tourniquet** on the forearm, It will likewise dwell for 2 minutes under occlusion before tourniquet release. This tourniquet method for lidocaine is known to significantly improve its efficacy in preventing injection pain
  Interventions: Drug: Lidocaine, a local anaesthetic.

INTERVENTIONS:
Drug: Lidocaine, a local anaesthetic. — it will be given as a pretreatment prior to injection of propofol, with a tourniquet applied.
  Arms: Lidocaine
Drug: Parecoxib 40mg — atients in this group will receive IV parecoxib 40 mg (the standard full dose for an adult) diluted to a total volume of 5 mL with normal saline.
  Arms: Parecoxib

SUMMARY:
Propofol is the most popular IV anaesthetic agent used for induction, however one of its known side effects is causing pain on injection, the gold standard method in preventing this pain is using lidocaine prior to injecting propofol. multiple drugs have been investigated to reduce the aforementioned pain, however there has been no study comparing lidocaine to parecoxib, an NSAID.

DETAILED DESCRIPTION:
Propofol is the most popular drug used for induction of anaesthesia. without prophylaxis, 60 to 70% of patients are affected by pain upon injection, with varying degrees of severity. The specific mechanism triggering pain is undetermined, but it is thought to be due to triggering of kallikrein-kinin cascade when it is injected.

Many strategies have been investigated to reduce the severity of this pain, with the most effective being the use of a large vein to deliver the drug, combined with pretreatment using lidocaine with venous occlusion to allow it to anaesthetize the vein locally. This approach has been shown in a large meta-analysis to be the gold standard for reducing pain caused by propofol injection, achieving up to an 80% reduction in incidence. However, this method is not widely used clinically, probably due to the extra time required to anaesthetize the vein and applying a tourniquet. On the other hand, using lidocaine as a pre- treatment or mixed with propofol has been shown to reduce pain on injection.

Multiple other agents have been investigated with the aim of preventing the pain caused by propofol injection, such as opioids and ketamine. Non-steroidal Anti inflammatory Drugs (NSAIDs) have also been studied, with the rationale that reducing prostaglandin production caused by the suggested cascade above. These medications are usually used as part of the multimodal analgesia delivered to the patient to prevent intraoperative and postoperative pain, if given prior to propofol, they may have the added benefit of reducing the pain caused by injecting propofol.

Parecoxib, a selective COX-2 inhibitor in the NSAIDs class, has been investigated recently in trails to prevent pain on injection caused by propofol, where a prospective Randomised controlled trial showed that a dose of 40 mg was effective in reducing the frequency and the severity of the pain, where the incidence of pain was only 26%, compared to 58% in the placebo group. Furthermore non of the patients in this group reported moderate or severe pain. In the same study, a 20 mg Dose was only shown to reduce the severity of pain and not the incidence.

The Investigators propose this study to compare the two interventions as no previous study has investigated them in the same setting.

Objective of the study.

To compare the efficacy of intravenous parecoxib versus lidocaine in reducing pain during propofol injection in adult ASA I-II patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years
* ASA grading I-II
* Patients undergoing elective surgical procedures across all surgical specialties.
* Can speak Arabic or English

Exclusion Criteria:

* Difficulty in communicating.
* Liver Cirrhosis patients
* Renal failure or creatinine clearance (CrCl) ≤ 10umol/L,
* Known Lidocaine, parecoxib and/or propofol allergy.
* patients who are not using propofol for an induction.
* Any known contraindication to propofol, parecoxib or lidocaine. (this will include renal failure or cirrhosis of the liver as noted above)
* Patients refusing to be involved in the study.
* ASA(American society of anaesthesia) grading 3-6.
* Any patient that IV access cannot be established in the dorsum of the hand.
* Pregnant women.
* Patients with chronic pain disorders.
* Patients who received any form of analgesia within the last hour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of pain on injecting propofol after receiving the treatment assigned. | immediately after injection of 50 mg of propofol.

SECONDARY OUTCOMES:
Severity of pain. | immediately after injection of propofol.
  Measured Via Visual analogue scale for pain. The patient will be given 50 mg of propofol and asked if there is any pain, and the severity of the pain. The severity of pain will be graded on the scale between 1 and 10, 10 being the most severe in the scale, and 1 is the minimal pain experienced.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker BJ, Neal JM, Mulroy MF, Humsi JA, Bittner RC, McDonald SB. Lidocaine pretreatment with tourniquet versus lidocaine-propofol admixture for attenuating propofol injection pain: a randomized controlled trial. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):41-5. doi: 10.1097/AAP.0b013e31820306da. PMID 21455088
- [Background] Tan CH, Onsiong MK. Pain on injection of propofol. Anaesthesia. 1998 May;53(5):468-76. doi: 10.1046/j.1365-2044.1998.00405.x. PMID 9659020
- [Background] Ghai B, Makkar JK, Bala I, Wig J. Effect of parecoxib pretreatment and venous occlusion on propofol injection pain: a prospective, randomized, double-blinded, placebo-controlled study. J Clin Anesth. 2010 Mar;22(2):88-92. doi: 10.1016/j.jclinane.2009.03.011. PMID 20304348
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529